CLINICAL TRIAL: NCT06610526
Title: An Interventional, Multicentre, Phase IV, Single-Arm, Open-Label Study to Investigate the Efficacy and Safety of Dapagliflozin in Chinese Adult Patients With Chronic Kidney Disease
Brief Title: A Study of Dapagliflozin in Chinese Adult Patients With Chronic Kidney Disease
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D169AC00008
Record Dates: First submitted 2024-08-20; First posted 2024-09-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg once daily
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin by oral administration

SUMMARY:
The purpose of this study is to describe the efficacy and safety information with dapagliflozin in Chinese patients with chronic kidney disease.

DETAILED DESCRIPTION:
This is an interventional, multicentre, Phase IV, single-arm, open-label study to investigate the efficacy and safety of dapagliflozin to prevent the progression of chronic kidney disease in Chinese adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study specific procedures
* Chinese Female or male aged ≥ 18 years at the time of consent
* eGFR ≥ 25 and ≤ 75 mL/min/1.73m2 (CKD-EPI Formula) at visit 1
* Evidence of increased albuminuria 3 months or more before visit 1 and UACR ≥ 200 and ≤ 5000 mg/g at visit 1
* Stable, and for the patient maximum tolerated labelled daily dose, treatment with ACE-I or ARB for at least 4 weeks before visit 1, if not medically contraindicated

Exclusion Criteria:

* Autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis or anti-neutrophil cytoplasmic antibodies-associated vasculitis
* Receiving cytotoxic therapy, immunosuppressive therapy or other immunotherapy for primary or secondary renal disease within 6 months prior to enrolment
* History of organ transplantation
* Receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor
* T1DM
* New York Heart Association class IV Congestive Heart Failure at the time of enrolment
* MI, unstable angina, stroke or TIA within 12 weeks prior to enrolment
* Coronary revascularization (PCI or CABG) or valvular repair/replacement within 12 weeks prior to enrolment
* Any condition outside the renal and CV disease area, such as but not limited to malignancy, with a life expectancy of less than 2 years based on investigator´s clinical judgement
* Active malignancy requiring treatment at the time of visit 1 (with the exception of successfully treated basal cell or treated squamous cell carcinoma)
* Hepatic impairment (AST or ALT > 3 × ULN; or total bilirubin > 2 × ULN at time of enrolment). An solated increase in bilirubin in patients with known Gilbert's syndrome is not a reason for exclusion
* Known blood-borne diseases
* Women of child-bearing potential (ie, those who are not chemically or surgically sterilised or who are not post-menopausal) who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator, from the time of signing the informed consent throughout the study and 4 weeks thereafter, OR women who have a positive pregnancy test at enrolment OR women who are breast-feeding
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca personnel and/or site personnel)
* Previous enrolled in the present study
* Participation in another clinical study with a study intervention during the last month prior to enrolment
* Inability of the patient, in the opinion of the investigator, to understand and/or comply with study intervention, procedures and/or follow-up OR any conditions that, in the opinion of the investigator, may render the patient unable to complete the study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of any of the components of the composite: 50% sustained decline in eGFR or Reaching ESRD or CV Death or Renal Death. | Up to a median follow-up time of 24 months
  Data is reported as descriptive statistics.

SECONDARY OUTCOMES:
Percentage change in UACR from baseline | Up to a median follow-up time of 24 months
  Data is reported as descriptive statistics.
Time to the first occurrence of any of the components of the composite: ≥ 50% sustained decline in eGFR or Reaching ESRD or Renal death | Up to a median follow-up time of 24 months
  Data is reported as descriptive statistics.
Time to the first occurrence of either of the components of the composite: CV death or Hospitalization for heart failure | Up to a median follow-up time of 24 months
  Data is reported as descriptive statistics.
Time to death from any cause | Up to a median follow-up time of 24 months
  Data is reported as descriptive statistics.
Measure the change in eGFR over time from baseline to the end of treatment and from first on treatment measurement to end of treatment | Up to a median follow-up time of 24 months
  Data is reported as descriptive statistics.
To describe the safety profile in Chinese adult patients with CKD treated with dapagliflozin: SAE, DAEs, and clinical chemistry/haematology parameters | From the administration of study intervention throughout the study until and including the patient's last visit, up to a median follow-up time of 24 months
  * The number and percent of subjects with SAE and DAE, and the total number of SAE and DAEs will be provided.
  * The result and the change from baseline of each clinical chemistry/haematology tests will be summarized at each scheduled visit using summary statistics based on the FAS.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Dongguan
  - Research Site, Foshan
  - Research Site, Fuyang
  - Research Site, Fuzhou
  - Research Site, Ganzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hengyang
  - Research Site, Huaian
  - Research Site, Huizhou
  - Research Site, Jilin
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Lanzhou
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Suzhou
  - Research Site, Taian
  - Research Site, Tianjin
  - Research Site, Wuhu
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xiamen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/